CLINICAL TRIAL: NCT06811038
Title: Providing Nicotine Replacement Therapy to Enhance the Efficacy of a Smoking Cessation Smartphone App for Hispanic Adults
Brief Title: iCanQuit Smoking Cessation Among Hispanic Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG1124868; NCI-2024-10014 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20697 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA298383 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices; Nicotine; Interviews as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To assure blinding, random assignments will be concealed from participants and researchers throughout the trial. Follow-up data will be collected by our survey research unit that will be blind to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm I (iCanQuit application) (Experimental): Participants receive access to the iCanQuit smartphone application for 12 months and complete personalized quit plans with education regarding managing urges, motivation, and relapse prevention, on-demand help with tracking of daily cigarette consumption, and monitoring of urges passed without smoking.
  Interventions: Device: iCanQuit Smartphone App Smoking Cessation Program; Other: Survey Administration; Other: Interview
- Arm II (iCanQuit application and NRT) (Experimental): Participants receive access to the iCanQuit smartphone application for 12 months and complete personalized quit plans with education regarding managing urges, motivation, and relapse prevention, on-demand help with tracking of daily cigarette consumption, and monitoring of urges passed without smoking. Participants also receive NRT patch(es) and gum to use per the usage instructions tailored to the participants' baseline smoking levels. In addition, participants receive daily push notifications with NRT dosage and refill reminders for 12 months.
  Interventions: Device: iCanQuit Smartphone App Smoking Cessation Program; Drug: Nicotine Gum; Drug: Nicotine Patch; Drug: Nicotine Lozenge; Other: Survey Administration; Other: Interview

INTERVENTIONS:
Device: iCanQuit Smartphone App Smoking Cessation Program — Receive access to iCanQuit app, with daily push notifications
  Other Names: iCanQuit
Drug: Nicotine Gum — Receive nicotine replacement therapy gum
  Other Names: Nicorette; Nicotine Polacrilex gum
  Arms: Arm II (iCanQuit application and NRT)
Drug: Nicotine Patch — Receive nicotine replacement therapy patch(es)
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
  Arms: Arm II (iCanQuit application and NRT)
Drug: Nicotine Lozenge — Receive nicotine replacement therapy lozenge(s)
  Other Names: Nicorette; mini lozenge; Nicotine Polacrilex lozenge
  Arms: Arm II (iCanQuit application and NRT)
Other: Survey Administration — Ancillary studies
Other: Interview — Ancillary studies

SUMMARY:
This phase III trial compares a smartphone application with or without nicotine replacement therapy in improving smoking cessation among Hispanic adults who would like to quit smoking. The iCanQuit smartphone application focuses on skills for managing urges, motivation, and relapse prevention with personalized quit plans. Nicotine replacement therapy works by giving small, steady doses of nicotine to help stop cravings and relieve symptoms that occur when a person is trying to quit smoking without any of the other harmful chemicals found in tobacco products.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive access to the iCanQuit smartphone application for 12 months and complete personalized quit plans with education regarding managing urges, motivation, and relapse prevention, on-demand help with tracking of daily cigarette consumption, and monitoring of urges passed without smoking.

ARM II: Participants receive access to the iCanQuit smartphone application for 12 months and complete personalized quit plans with education regarding managing urges, motivation, and relapse prevention, on-demand help with tracking of daily cigarette consumption, and monitoring of urges passed without smoking. Participants also receive NRT patch(es) and gum or lozenges to use per the usage instructions tailored to the participants' baseline smoking levels. In addition, participants receive daily push notifications with NRT dosage and refill reminders for 12 months.

After completion of study intervention, patients may be followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic ethnicity
* Age 18 and older
* Smoking at least one cigarette per day in the past 30 days
* Want to quit smoking within 30 days
* Interest in learning skills to quit smoking
* Willing to be randomly assigned
* United States (US) or Puerto Rico (PR) residency for the next twelve months
* Have daily access to their own Android or iPhone smartphone
* Ability to download a smartphone application (app)
* Proficiency in English or Spanish
* Not currently (i.e., within past 30 days) using other smoking cessation interventions
* Willing to consider using NRT
* No previous use of iCanQuit
* No household or family member participating
* Willingness to complete follow-up assessments at the 3-, 6-, and 12-month follow-ups
* Providing email, phone number(s), and mailing address

Exclusion Criteria:

* NRT CONTRAINDICATION: Heart attack in the last 2 months
* NRT CONTRAINDICATION: Stroke in the last 6 months
* NRT CONTRAINDICATION: Diagnosed arrhythmia or tachycardia
* NRT CONTRAINDICATION: Uncontrolled hypertension
* NRT CONTRAINDICATION: Currently using warfarin
* NRT CONTRAINDICATION: Pregnant or breastfeeding, or plans to become pregnant during the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 854 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
30-day point prevalence abstinence (PPA) | At 12 months post randomization
  The comparison will use a logistic regression model, following standard intent-to-treat analysis for smoking cessation trials, will be employed, coding all missing outcomes as smoking. The model will adjust for stratification factors and baseline factors that are both imbalanced after randomization and significantly related to the outcome.

SECONDARY OUTCOMES:
30-day PPA | At 3 and 6 months post randomization
24 hour PPA | At 3, 6 and 12 months post randomization
7 day PPA | At 3, 6 and 12 months post randomization
Cost per quitter | At 12 months post randomization
  Standard methods for estimating cost-effectiveness in smoking cessation interventions will be used. The incremental cost-per-quitter will be estimated as the difference in total cost of delivering the two interventions divided by the difference in the number of 30-day abstinent participants at 12 months.
Cost per life year gained | At 12 months post randomization
  Standard methods for estimating cost-effectiveness in smoking cessation interventions will be used. To compare iCanQuit with iCanQuit plus NRT in terms of life years gained, researchers will calculate the cost per life year gained.
Cost per quality-adjusted life year (QALY) gained | At 12 months post randomization
  Standard methods for estimating cost-effectiveness in smoking cessation interventions will be used. Will estimate cost-per-QALY gained.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The trial results data will be published on ClinicalTrials.gov at the time of study completion. The de-identified scientific data will be made available to other users no later than the time of publication of the primary outcomes, or at the end of the performance period, whichever comes first. The de-identified scientific data will be made available as public use data to the research community in openICPSR. Members of the research community using this data must register with ICPSR and agree to the Terms of Use, which include limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, requiring immediate reporting of any disclosure of participant identity, and requiring users agree not to share or redistribute any data downloads. No PII or PHI data will be shared or available for secondary use. The de-identified data deposited in openICPSR will be available to the research community in perpetuity.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The trial results data will be published on ClinicalTrials.gov at the time of study completion. The de-identified scientific data will be made available to other users no later than the time of publication of the primary outcomes, or at the end of the performance period, whichever comes first. The de-identified data deposited in openICPSR will be available to the research community in perpetuity.
Access Criteria: The de-identified scientific data will be made available as public use data to the research community in openICPSR. Members of the research community using this data must register with ICPSR and agree to the Terms of Use, which include limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, requiring immediate reporting of any disclosure of participant identity, and requiring users agree not to share or redistribute any data downloads. No PII or PHI data will be shared or available for secondary use.